CLINICAL TRIAL: NCT06531109
Title: PRESTO - Characterization and Clinical Outcomes of Alopecia Aerata (AA) Patients Treated With Ritlecitinib in a Real-world (RW) Cohort: A Multinational, Prospective Observational Study.
Brief Title: Characterization And Clinical Outcomes of AA Patients Treated With Ritlecitinib
Acronym: PRESTO
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7981105; NCT06531109 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-07-11; First posted 2024-07-31 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alopecia Areata (AA) patients treated with ritlecitinib
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Ritlecitinib — As provided in the real world practice.

SUMMARY:
Alopecia areata (AA) is a chronic relapsing autoimmune disease characterized by nonscarring hair loss affecting children, adolescents, and adults across all ages, races, and genders. AA primarily affects the scalp; however, it also can affect nails, eyelashes, eyebrows, and other hair follicles on the patient's body. The 3 main types of AA are:

* Patchy alopecia (PA), as seen in 90% of clinical diagnoses
* Alopecia totalis (AT), that affects all scalp hair
* Alopecia universalis (AU), involving all scalp, face, and body hair Dermatologist preferences for utility and order of skin-directed therapies to treat AA vary widely, with treatment choices based on various factors such as patients' age, disease duration and severity (Meah et al., 2020).

Ritlecitinib is a bioavailable small molecule that irreversibly binds to Janus kinase-3 (JAK3) and Tyrosine kinase Expressed in the hepatocellular Carcinoma kinase family (TEC). Ritlecitinib 50 mg once daily was approved by the FDA 23 June 2023 and EMA 20 July 2023 for the treatment of severe alopecia areata in adults and adolescents 12 years of age and older. In Japan, ritlecitinib was approved on 26 June 2023 for the treatment of alopecia areata (limited to intractable cases involving widespread hair loss). Additional countries have since approved ritlecitinib. Those approvals are based on the results of the ritlecitinib pivotal phase 2b/3 study (ALLEGRO 2b/3) which examined efficacy and safety of ritlecitinib in AA patients globally.

Despite positive results from the ALLEGRO program, there is still lack of evidence on ritlecitinib patients' characteristics and clinical outcomes in routine clinical practice. The investigators will evaluate patient and disease characteristics, treatment patterns, and clinical and patient-reported outcomes among patients with AA who are receiving ritlecitinib.

The aim of this study is to measure effectiveness of ritlecitinib in a real-world setting. Ritlecitinib will be prescribed to patients according to the approved product label. Treatment will be guided by clinical judgement of the treating physician ie, study investigators, according to standard of care, independently of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged >12 years at baseline.
2. Patients with diagnosis of alopecia areata confirmed by a certified dermatologist, who are prescribed ritlecitinib as per the product label independently of the decision to enroll a patient in this study.
3. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study. Following receipt of oral and written information about the trial, the adolescent (depending on local institutional review board/independent ethics committee requirements) must provide assent, and one or both (according to local regulations) parents or guardians of the child must provide signed informed consent before any study-related activity is carried out.
4. Patients, who in the opinion of the investigator, are willing and able to comply with regular clinic visits as per standard practice at the site and agree to complete PRO questionnaires and other patient completed questions.

Exclusion Criteria:

1. Diagnosed with other types of alopecia or other diseases that can cause hair loss (including, but not limited to known androgenetic alopecia, traction and scarring alopecia, telogen effluvium).
2. Diagnosed with other scalp diseases that may impact AA assessment (e.g., scalp psoriasis, dermatitis, etc.) or other active systemic diseases that may cause hair loss (e.g., lupus erythematosus, thyroiditis, systemic sclerosis, lichen planus, etc.). that could interfere with assessment of hair loss/regrowth.
3. Patients previously treated with ritlecitinib or other JAK inhibitors.
4. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population eligible for enrollment includes any adult and adolescent patients aged ≥12 years diagnosed with AA who receive at least one dose of ritlecitinib and satisfy the inclusion and exclusion criteria. The study will be open for enrollment for approximately 12 months after the first patient has been enrolled. Depending on the observed enrollment rate, the enrollment period and number of sites may be reassessed and revised during the study. It will be allowed to enroll patients with previous use of topical JAK inhibitors only if there was at least a 4-week wash-out period prior to Baseline Visit
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in Severity of Alopecia Tool (SALT) score at week 24 | 24 weeks from initiation of the treatment
  SALT score is used to calculate the severity of alopecia areata. Physician calculate it by summing the percentage of hair loss in different regions of scalp.

SECONDARY OUTCOMES:
Demographic characteristic of participants: Age, sex, race, ethnicity, socio-economic status, area of residence, smoking status | Baseline
  Number/percentage of patients by age, sex, race, ethnicity, socio-economic status, area of residence, smoking status. Race and ethnicity variables will only be collected in participating countries where it is allowed.
Demographic Characteristic of Participants: Date of Initial AA diagnosis | Baseline
Demographic Characteristics of participants: Duration of AA since diagnosis | Baseline
Demographic characteristics of participants: Duration of current AA Episode | Baseline
Demographic Characteristic of Participants: Predominant AA phenotype | Baseline
  Predominant AA phenotype (eg, patchy; ophiasis; AT; AU, etc
Clinical Characteristics of participants: Severity of Alopecia Tool (SALT) Score | Baseline
  SALT score is used to calculate the severity of alopecia areata.
Clinical characteristics of participants: Eyelash Assessment (ELA) score | Baseline
  ELA score is used to calculate the severity of the involvement of eyelashes.
Clinical Characteristics of participants: Eyebrow Assessment (EBA) Score | Baseline
  EBA score is used to calculate the severity of the involvement of eyebrows
Clinical Characteristics of participants: number of affected nails | Baseline
Clinical Characteristics of participants: Presence of Beard involvement | Baseline
  Determine whether the beard is affected or not.
AA treatment history of participants: number of patients with prior AA treatments | Baseline
AA treatment history of participants: prior AA treatment class and route | Baseline
AA treatment history of participants: duration of prior therapy / frequency | baseline
AA treatment history of the participants: total number of prior AA treatments | Baseline
RW effectiveness of ritlecitinib: proportion of patients with <20 in SALT score | week 24, 48, 72 and 96
  decrease in SALT score is the indicator of effectiveness.
RW effectiveness of ritlecitinib: Proportion of patients with <10 | week 24, 48, 72 and 96
  Decrease in SALT score is the indicator of effectiveness
RW effectiveness of ritlecitinib: Change from baseline in SALT score | week 24, 48, 72 and 96
  Decrease in SALT score is the indicator of effectiveness
RW effectiveness of ritlecitinib: proportion of patient with improvement from abnormal baseline in Eyebrow Assessment score (EBA) | Week 24, 48, 72 and 96
  Improvement in EBA score will indicate ritlecitinib effectiveness in eyebrow involvement.
RW effectiveness of ritlecitinib: proportion of patient with improvement from abnormal baseline in Eyelashes Assessment Score (ELA) | Week 24, 48, 72 and 96
  Improvement in ELA score will indicate ritlecitinib effectiveness in eyebrow involvement.
RW effectiveness of ritlecitinib: proportion of patients with improvement from abnormal baseline in beard assessment and nail involvement | week 24, 48, 72 and 96
Patient reported outcome: Evaluate ritlecitinib treatment satisfaction | week 24, 48, 72 and 96
  Patient-reported satisfaction (P-sat) Response (defined as slightly, moderately, or very satisfied) at 24, 48, 72 and 96 weeks
Patient reported outcome: Evaluate impression of hair growth | week 24, 48, 72 and 96
  Patient Global Impression of Change (PGI-C) Response (defined as a score of moderate to severe), at 24, 48, 72 and 96 weeks
Evaluate impact of ritlecitinib: Patient reported quality of life | week 24, 48, 72 and 96
  Changes in AAPPO. · Improvement in hair loss AAPPO items 1-4, defined as a score of 0="no hair loss" or
  1=" little hair loss", among patients with a baseline score 2-4 indicating moderate-complete hair loss.
Evaluate impact of ritlecitinib: Patient reported quality of life | week 24, 48, 72 and 96
  Change from baseline in emotional symptoms (ES) and activity limitations (AL) subscores

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- United States (25):
  - C2 Research Center, Montgomery, Alabama
  - CENTER FOR DERMATOLOGY CLINICAL RESEARCH, Inc, Fremont, California
  - Rao Dermatology, Fresno, California
  - Cura Clinical Research, Oxnard, California
  - Southern California Clinical Research, Santa Ana, California
  - Dermatology of Boca, Boca Raton, Florida
  - Pediatric Skin Research,LLC, Coral Gables, Florida
  - Suncoast Skin Solutions, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Skin Research of South Florida LLC, Miami, Florida
  - Kindred Hair and Skin Center, Marriottsville, Maryland
  - Brigham & Women's Hospital/Harvard Medical School, Boston, Massachusetts
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Michigan Dermatology Institute, Waterford, Michigan
  - Twin Cities Dermatology Center, Minneapolis, Minnesota
  - Central Missouri Dermatology Research, Columbia, Missouri
  - Hickory Dermatology Research Center, Hickory, North Carolina
  - NW Dermatology Institute, Portland, Oregon
  - UPMC, Pittsburgh, Pennsylvania
  - Goodlettsville Dermatology Research, Goodlettsville, Tennessee
  - Epiphany Dermatology, Southlake, Texas
  - Raven Clinical Reseach, Fairfax, Virginia
  - Raven Clinical Reseach, McLean, Virginia
  - Frontier Dermatology, Mill Creek, Washington
  - Raven Clinical Reseach, Burlington, Wisconsin
- China (6):
  - Beijing Tongren Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Dermatology Hospital of Southern Medical University, Guangzhou
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Shanghai Skin Disease Hospital, Shanghai
- France (3):
  - Ch Victor Dupouy, Argenteuil
  - CHU de CAEN, Caen
  - Rouen University Hospital, Rouen
- Japan (8):
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Nagomi Dermatology Clinic, Ebina, Kanagawa
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo
- United Kingdom (6):
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucester, Gloucestershire
  - Royal United Hospital Bath, Bath
  - NHS Greater Glasgow and Clyde, Glasgow
  - Whipps Cross (Barts Health), London
  - London North West University Healthcare Trust, London
  - Chelsea and Westminster NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981105